CLINICAL TRIAL: NCT01265927
Title: A Phase I Study Inhibiting Telomerase to Reverse Trastuzumab Resistance in HER2+ Breast Cancer
Brief Title: A Study Inhibiting Telomerase to Reverse Trastuzumab Resistance in HER2+ Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Breast Cancer Research Foundation (Other); Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0314; 1010-05 (Other: IRB-02)
Record Dates: First submitted 2010-12-03; First posted 2010-12-23 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Breast Tumors; Cancer of Breast; Cancer of the Breast; Genes, HER-2; Genes, HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; imetelstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GRN163L + Trastuzumab (Experimental)
  Interventions: Drug: GRN163L in combination with trastuzumab

INTERVENTIONS:
Drug: GRN163L in combination with trastuzumab — GRN163L will be administered in escalating dose cohorts on Day 1 of each 21-day cycle prior to trastuzumab infusion. Trastuzumab will be a administered day 1 of each 21-day cycle after GRN163L. There will be a 30 minute observation period between the end of the GRN163L infusion and the beginning of the trastuzumab infusion.
  Other Names: Imetelstat Sodium; Herceptin

SUMMARY:
A study to evaluate safety and biologic effects of giving GRN163L in combination with trastuzumab in patients diagnosed with HER2+ metastatic breast cancer that is resistant to therapy with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 years or older at the time of consent.
2. ECOG performance status of 0-2 within 21 days of study registration.
3. Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease. NOTE: locally recurrent disease must not be amenable to surgery or radiation with curative intent.
4. Measurable or evaluable disease according to RECIST v1.1 within 35 days prior to study registration.
5. Disease must be amenable to biopsy (image-guided or via direct visualization of superficial lesions) with minimal risk to the patient. NOTE: Patients with disease limited to the lung and/or pleura are excluded.
6. Disease must be HER2+ as defined by IHC 3+ or FISH ratio > 2.0.
7. Resistant to trastuzumab as defined as (1) progression within 12 months of completing adjuvant/neoadjuvant trastuzumab or (2) progression on trastuzumab administered for metastatic disease.
8. Prior treatment with lapatinib or investigational HER2 targeted therapies is allowed but not required. There are no limits on the number of regimens or other prior anti-HER2 therapies patients have received.
9. LVEF ≥ Lower Limit of Normal based on MUGA or ECHO within 35 days prior to study registration
10. Females of childbearing potential and males must be willing to use an effective method of contraception from the time consent is signed until 6 months after treatment discontinuation. Methods of contraception include hormonal birth control (oral contraceptives, patch, injection, vaginal ring or implant), two barrier methods of birth control, abstinence and/or other methods as determined by the treating physician.
11. Females of childbearing potential must have a negative pregnancy test within 14 days prior to registration for protocol therapy.

    NOTE: Females are considered of child bearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal (> 12 months since last menses).

    Laboratory values must be obtained within 21 days of study registration:
12. Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
13. Platelets ≥ 100 K/mm3
14. Hemoglobin (Hgb) ≥ 9.0 g/dL (may be transfused)
15. Serum creatinine < 3.0 mg/dL
16. Total Bilirubin ≤ 1.5 x ULN
17. AST/SGOT ≤ 2.5 x ULN. If liver metastases is present, AST ≤ 5 x ULN
18. ALT, SGPT ≤ 2.5 x ULN. If liver metastases is present, ALT ≤ 5 x ULN

    Exclusion Criteria:
19. No Investigational therapy within 4 weeks of study registration
20. No hormonal therapy within 2 weeks of study registration
21. No cytotoxic chemotherapy within 2 weeks of study registration.
22. No prior treatment with GRN163L
23. No prior history of severe reaction to trastuzumab, as determined by the treating physician.
24. No history of clinically significant cardiac dysfunction, including:

    Current uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg), or unstable angina History of symptomatic CHF (Grade >3 by NCI CTCAE or Class >II by NYHA criteria [see Appendix IV]) or serious cardiac arrhythmia requiring treatment within 12 months of study registration, with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia History of myocardial infarction within 6 months of study registration
25. No history of cerebrovascular accident within 12 months of study registration
26. No active CNS metastases. Patients with previously treated CNS metastases who do not require chronic steroids or anticonvulsants are eligible.
27. Prior radiation therapy must not have involved > 25% of bone marrow due to potential myelosuppression with GRN163L. See bone marrow chart in Appendix III

    NOTE: Radiation therapy within 2 weeks of study registration is not allowed.
28. Females must not be breastfeeding.
29. No clinically significant active infection, as determined by the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determine the dose-limiting toxicity of GRN163L in combination with trastuzumab in patients with refractory HER2+ metastatic disease | End of Study

SECONDARY OUTCOMES:
Measure the concentration of trastuzumab and GRN163L from blood samples immediately before and after infusion on day 1, weekly during cycle 1, and immediately prior to cycle 2 | Until cycle 2
  PK data will be described using means, standard deviations, medians, minimums and maximums.
Tumor biopsy and bone marrow aspirate assayed for telomerase activity prior to treatment and immediately prior to planned cycle 2 | Until cycle 2
  Telomerase activity data will be described using means, standard deviations, medians, minimums and maximums.
Flow cytometry to compare cell cycle distribution in tumor and bone marrow prior to treatment and immediately prior to cycle 2. | Until cycle 2
  Marrow (and tumor when sufficient sample is available) will be analyzed via flow cytometry to determine cell distribution. Percentage of cells at each cycle will be described using means, standard deviations, medians, minimums and maximums.
Tumor samples analyzed for activation of HER2 family signaling protein activation (phosphorylation) status prior to treatment and immediately prior to cycle 2. | Until cycle 2
  HER2 family signaling protein activation will be described using means, standard deviations, medians, minimums and maximums.
Determine objective response rate (ORR) and progression free survival (PFS) of GRN163L in combination with trastuzumab in this patient population | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States